CLINICAL TRIAL: NCT00002593
Title: Phase III Randomized Trial of 5-FU/Leucovorin/Levamisole Versus 5-FU Continuous Infusion/Levamisole as Adjuvant Therapy for High-Risk Resectable Colon Cancer
Brief Title: S9415 Chemotherapy in Patients With Stage II or III Colon Cancer That Has Been Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000063773; SWOG-9415 (Other: SWOG); CLB-9498 (Other: CALGB); INT-0153 (Other: NCI); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Levamisole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-FU/Leucovorin/Levamisole (Active Comparator): levamisole hydrochloride: 50 mg every 8 hours x 3 days, PO, repeat every 14 days for 6 months; leucovorin calcium: 20 mg/m^2/day, IV, Days 1-5 of each cycle; 5-fluorouracil: 425 mg/m^2/day, IV, Days 1-5 of each cycle;
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: levamisole hydrochloride
- Infusional 5-FU + Levamisole (Active Comparator): levamisole hydrochloride : 50 mg every 8 hours x 3 days, PO, repeat every 14 days for 6 months; 5-fluorouracil: 250 mg/m^2/day, continuous infusion, daily for 56 days x 3 cycles of 8 weeks.
  Interventions: Drug: fluorouracil; Drug: levamisole hydrochloride

INTERVENTIONS:
Drug: fluorouracil — Given IV as described in Arm Description
  Other Names: 5-fluorouracil; 5-FU; NSC-19893
Drug: leucovorin calcium — Given IV as described in Arm description.
  Other Names: Leucovorin; Folinic acid; NSC-3590
  Arms: 5-FU/Leucovorin/Levamisole
Drug: levamisole hydrochloride — Given as described in arm description
  Other Names: Levamisole; NSC-177023

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy given in different ways in treating patients with surgically removed stage II or stage III colon cancer at high risk of recurrence.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall and disease free survival in patients with completely resected stage II or III colon cancer randomized to adjuvant chemotherapy with bolus fluorouracil and leucovorin calcium with levamisole vs continuous infusion fluorouracil with levamisole.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, T stage (T1 vs T2 vs T3 vs T4a), N stage (N0 vs N1 vs N2-3), and time from surgery until registration (21-28 vs 29-35 days). Patients are randomized to one of two treatment arms. Arm I: Patients receive leucovorin calcium IV immediately followed by fluorouracil IV on days 1 through 5 of weeks 1, 5, 9, 14, 19, and 24, and oral levamisole 3 times a day for 3 days on days 1-3. Courses repeat every 2 weeks for 6 months. Arm II: Patients receive levamisole as in arm I plus fluorouracil by continuous IV infusion for 8 weeks. Treatment with fluorouracil repeats every 10 weeks for 3 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed at 9 months and 12 months, then every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,500 patients will be accrued for the study over approximately 5.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven resectable stage II or III adenocarcinoma of the colon Caudal margin of the primary tumor must lie above the peritoneal reflection Must have pathologic confirmation of either N1-3 (stage III), or if N0, must have T3-T4 (stage II) with bowel obstruction or perforation Obstruction documented as: At least 75% colon or small bowel obstruction on x-ray and/or endoscopy Significant bowel dilatation surgically documented Significant obstruction described in the pathology report Perforation documented by gross operative/pathologic evidence of a colon wall defect with associated abscess or peritonitis Complete en bloc resection by laparotomy required No laparoscopic colectomy without prior surgery on protocol SWOG-9411 No gross or microscopic residual disease No distant peritoneal metastases (stage IV) even if grossly resectable No requirement to open the pelvic peritoneum to define the extent of disease No extrapelvic nodal metastasis unless resected en bloc with the primary tumor No distant metastases No other diagnosis of stage II-III colon cancer within the past 5 years May have undergone complete surgical resection at least 5 years prior to study Completely resected prior or synchronous stage 0-I colon cancer eligible

PATIENT CHARACTERISTICS: Age: Adult Performance status: SWOG 0-2 Hematopoietic: WBC (white blood cell) at least 3,500/mm3 Platelet count at least within the lower limit of normal Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST (angiotensin sensitivity test) no greater than 2 times ULN Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine no greater than 2 times ULN Other: No organic brain syndrome, Alzheimer's disease, or other altered mental status No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Adequately treated carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior fluorouracil or other chemotherapy for cancer No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior or concurrent radiotherapy for cancer Surgery: Complete en bloc resection required (see Disease Characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1135 (Actual)
Dates: Start 1994-12; Primary Completion 1999-12 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Compare effectiveness of bolus 5-FU, leucovorin, levamisole vs continuous infusion 5-FU, levamisole as adjuvant therapy for patients with colon cancer, measured in overall survival | At death

SECONDARY OUTCOMES:
Disease free survival | Until progression

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Poplin, MD, Study Chair — Rutgers Cancer Institute of New Jersey; Robert J. Mayer, MD, FACP, Study Chair — Dana-Farber Cancer Institute; Daniel G. Haller, MD, Study Chair — Abramson Cancer Center at Penn Medicine; Richard M. Goldberg, MD, Study Chair — Mayo Clinic
Locations (60):
- United States (57):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada
- Veterans Affairs Medical Center - San Juan, San Juan, Puerto Rico
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Background] Yothers G, Sargent DJ, Wolmark N, Goldberg RM, O'Connell MJ, Benedetti JK, Saltz LB, Dignam JJ, Blackstock AW; ACCENT Collaborative Group. Outcomes among black patients with stage II and III colon cancer receiving chemotherapy: an analysis of ACCENT adjuvant trials. J Natl Cancer Inst. 2011 Oct 19;103(20):1498-506. doi: 10.1093/jnci/djr310. Epub 2011 Oct 12. PMID 21997132
- [Result] Poplin EA, Benedetti JK, Estes NC, Haller DG, Mayer RJ, Goldberg RM, Weiss GR, Rivkin SE, Macdonald JS. Phase III Southwest Oncology Group 9415/Intergroup 0153 randomized trial of fluorouracil, leucovorin, and levamisole versus fluorouracil continuous infusion and levamisole for adjuvant treatment of stage III and high-risk stage II colon cancer. J Clin Oncol. 2005 Mar 20;23(9):1819-25. doi: 10.1200/JCO.2005.04.169. PMID 15774775
- [Result] Poplin E, Benedetti J, Estes N, et al.: Phase III randomized trial of bolus 5-FU/leucovorin/levamisole versus 5-FU continuous infusion/levamisole as adjuvant therapy for high risk colon cancer (SWOG 9415/INT-0153). [Abstract] Proceedings of the American Society of Clinical Oncology 19: A931, 2000.
- [Result] Leichman CG, Poplin E, Zalupski M, et al.: A pilot trial of infusion 5-fluorouracil with levamisole as adjuvant therapy for stage III colon cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 14: A-460, 196, 1995.